CLINICAL TRIAL: NCT04946630
Title: A Single Site, Open Label, 4-inhalation Session, Explorative Clinical Investigation to Investigate the Ability of PreciseInhale to Direct Regional Lung Targeting and Reduce the Degree of Throat Deposition and Subsequent Gastrointestinal Absorption in Healthy Volunteers After Inhalation of Test Drug Substances Via the PreciseInhale System
Brief Title: Explorative Clinical Investigation to Investigate the Ability of PreciseInhale to Direct Regional Lung Targeting and Reduce the Degree of Throat Deposition and Subsequent Gastrointestinal Absorption in Healthy Volunteers After Inhalation of Test Drug Substances Via the PreciseInhale System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inhalation Sciences Sweden AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); PlantVision AB (Unknown); Pharm-Analyt Labor GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLIN01-PI
Record Dates: First submitted 2021-06-04; First posted 2021-07-01 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: The 4 treatment periods will include 4 inhalation sessions. The 12 included subjects will participate in all 4 treatment periods and the same order of treatment periods will be followed for all included subjects. There will be a wash-out period of at least 1 week between treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Seretide Evohaler forte according to SmPc (Experimental): Single dose inhalation of fluticasone propionate/salmeterol 250 µg/25 µg administered via the Evohaler in accordance with instruction in the SmPC for Seretide Evohaler forte.
  Interventions: Other: Seretide Evohaler forte
- Whole lung exposure (Experimental): Single dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for whole lung exposure. The entire 300 mL aerosol volume produced by the single dose from the inhaler will be inhaled at a flow rate in accordance with instructions for the Evohaler.
  Interventions: Device: PreciseInhale; Other: Seretide Evohaler forte
- Alveolar bolus/ Breath hold exposures (Experimental): A subdivided dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for six repetitive 70 mL Alveolar bolus/ Breath hold exposures. Each 70 mL bolus will be extracted from a freshly generated volume of 300 mL aerosol produced by actuation of a single dose from the inhaler.
  Interventions: Device: PreciseInhale; Other: Seretide Evohaler forte
- Bronchial bolus/ Breath hold exposures (Experimental): A subdivided dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for six repetitive 70 mL Bronchial bolus/ Breath hold exposures. Each 70 mL bolus will be extracted from a freshly generated volume of 300 mL aerosol produced by actuation of a single dose from the inhaler.
  Interventions: Device: PreciseInhale; Other: Seretide Evohaler forte

INTERVENTIONS:
Device: PreciseInhale — Three different settings of the medical device PreciseInhale will be used in the study; PreciseInhale Whole Lung Exposure, PreciseInhale Bronchial Bolus/Breath hold Exposure and PreciseInhale Alveolar Bolus/Breath hold Exposure.
  Arms: Alveolar bolus/ Breath hold exposures; Bronchial bolus/ Breath hold exposures; Whole lung exposure
Other: Seretide Evohaler forte — Single dose of Seretide Evohaler forte (fluticasone propionate/salmeterol 250 µg/25 µg) administered according to SmPc or via the PreciseInhale system.

SUMMARY:
This is a single site, open label, 4-inhalation sessions, explorative clinical investigation to investigate the ability of PreciseInhale to direct regional lung targeting and reduce the degree of throat deposition and subsequent gastrointestinal absorption of test drug substances in healthy volunteers after inhalation of test drug substances via the PreciseInhale system.

The study will include a screening visit, 8 consecutive treatment visits and a follow-up telephone call 3-5 days after the last inhalation session. There will be a screening period of up to 35 days and an at least 1-week washout between treatments.

DETAILED DESCRIPTION:
Intended use The PreciseInhale system is a benchtop aerosol generation and dispensation system set up for extracting aerosol from clinical inhalers. The PreciseInhale system is classified as a Class IIa device according to MDD Annex IX, Rule 11.

PreciseInhale is intended to administer test drug substances in precise doses by producing exact amounts of inhalable aerosols from a clinical inhaler.

Extraction of the aerosol and exposure to humans must comply with operator and test subject safety regulations and only conducted in accordance with permits from the Swedish Medical Products Agency (MPA) and Swedish Ethical Review Authority (SERA) if necessary.

Indication PreciseInhale is not intended to treat any specific condition that requires medical attention. The purpose of the clinical investigation is to prove that the principle of operation of PreciseInhale is useful for administration of aerosols to humans.

Methodology Screening (Visit 1) will take place from Day -35 to Day 1 and will include general health assessments and an eligibility check.

At Visits 2 to 9, subjects will be admitted to the research clinic on Day -1 and will remain at the research clinic for PK and safety assessments until at least 12 hours after a single dose fluticasone propionate/salmeterol 250/25 µg is administered on the morning of Day 1 (Visit 2, 4, 6 and 8). The subjects will be carefully monitored by clinical staff during and after dosing. Vital signs and ECG will be checked at pre-determined timepoints. There is immediate access to equipment and qualified staff in case of an emergency.

Fluticasone propionate/salmeterol will be administered to each subject via the Evohaler or the PreciseInhale system, in the morning of Day 1 of each treatment period.

The 4 treatment periods will include these 4 inhalation sessions (up to 5 minutes/per session):

1. Single dose inhalation of fluticasone propionate/salmeterol 250 µg/25 µg administered via the Evohaler in accordance with instruction in the SmPC for Seretide Evohaler forte.
2. Single dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for whole lung exposure. The entire 300 mL aerosol volume produced by the single dose from the inhaler will be inhaled at a flow rate in accordance with instructions for the Evohaler.
3. A subdivided dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for six repetitive 70 mL Alveolar bolus/ Breath hold exposures. Each 70 mL bolus will be extracted from a freshly generated volume of 300 mL aerosol produced by actuation of a single dose from the inhaler.
4. A subdivided dose of fluticasone propionate/salmeterol 250 µg/25 µg administered via the PreciseInhale system set up for six repetitive 70 mL Bronchial bolus/ Breath hold exposures. Each 70 mL bolus will be extracted from a freshly generated volume of 300 mL aerosol produced by actuation of a single dose from the inhaler.

Inhalations will be administered by trained study personnel and the subjects will receive inhalation training before each inhalation session.

Subjects will be served a light breakfast before each treatment administration. After 1 hour post dose, the meal intake is unrestricted within the meal selection available at the research clinic. Lunch, Snack, dinner and evening snack (optional) will be served approximately 4, 6, 9 and 12 hours post-dose, respectively. Fluids will be restricted 1 hour prior to dosing until 1 hour after dosing. An optional breakfast may be served in the morning of Day 2 before the subject leaves the clinic.

PK samples will be collected at 17 time points in each treatment period: pre-dose, 2, 4, 6, 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours after treatment.

The subjects will be discharged from the research clinic in the evening of Day 1 (12 hours post treatment) and return to the research clinic in the morning (Visits 3, 5, 7 and 9; 24 hours post treatment) of Day 2 for PK sampling (and follow up safety assessments on the last Day 2).

There will be a wash-out period of at least 1 week between treatments. A follow-up telephone call (Visit 10, end-of-study) will be made 3-5 days after the last inhalation to follow-up on adverse events and device deficiencies.

A device user experience questionnaire will be completed by the study subject and PreciseInhale operator after all inhalation sessions with the PreciseInhale have been completed, i.e after the fourth inhalation session.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject aged ≥18 and ≤30 years inclusive.
3. Body Mass Index (BMI) ≥18 and ≤30 kg/m2 and weight ≥50 kg to ≤100 kg at screening.
4. Clinically normal medical history, physical findings, vital signs and laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

1. History of any clinically significant disease or disorder (including clinically significant disease affecting the respiratory tract, thoracic deformities affecting lung function and/or lung volumes, muscle diseases affecting lung function and/or lung volumes and any known mouth or nasal passage deformities) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within two weeks prior to the first inhalation with the investigational device, which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
3. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
4. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure > 140 mm Hg
   * Diastolic blood pressure > 90 mm Hg
   * Pulse < 40 or > 85 beats per minute
5. Former regular daily smoker.
6. Current smokers or users of nicotine products (including vaping/e-cigarettes). Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco, vaping) less than three times per week is allowed before the screening visit.
7. FVC or FEV1 outside of normal ranges (depending on subject's gender, height and age) at screening.
8. Female subjects who are pregnant or who are currently breast feeding.
9. Administration of a new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment with less than one month before the first inhalation session.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity (including pollen allergy), as judged by the Investigator.
11. History of hypersensitivity to drugs with a similar chemical structure or class to fluticasone or salmeterol, as judged by the Investigator.
12. Positive screen for drugs of abuse or alcohol at screening or on admission to the research unit prior to any of the inhalation sessions.
13. Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse.
14. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
15. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Cmax | From pre-dose to up to 24 hours post-dose.
  Maximum plasma concentration. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations of salmeterol and fluticasone propionate after administration of the test drug substances via the Evohaler or the PreciseInhale-device will be collected. Cmax (in plasma) will be compared for PreciseInhale versus inhalation directly from pMDI (Evohaler). Outcome measured in session 1-4.
AUC0-t | From pre-dose to up to 24 hours post-dose
  Area under the curve from time 0 to time t. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations of salmeterol and fluticasone propionate after administration of the test drug substances via the Evohaler or the PreciseInhale-device will be collected. AUC0-t (in plasma) will be compared for PreciseInhale versus inhalation directly from pMDI (Evohaler). AUC0-t (in plasma) will be compared for PreciseInhale versus inhalation directly from pMDI (Evohaler). Outcome measured in session 1-4.
Tmax | From pre-dose to up to 24 hours post-dose
  Time to Cmax. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations of salmeterol and fluticasone propionate after administration of the test drug substances via the Evohaler or the PreciseInhale-device will be collected.Tmax (in plasma) will be compared for PreciseInhale versus inhalation directly from pMDI (Evohaler). Outcome measured in session 1-4.
Inhaled and exhaled dose, fraction inhaled/exhaled dose | Collected post-dose at one occasion, approx. for 2 min
  Calculated inhaled dose (µg), dose in exhaled air (µg) and fraction inhaled/exhaled dose (analysed from PARI filter, data collected from inhalation sessions No. 2, 3 and 4). Outcome measured in session 2-4.
Inhaled and exhaled dose, fraction inhaled/exhaled dose | Collected post-dose at one occasion, approx. for 2 min
  Demonstrate that one inhaler aerosol dose from the pMDI can be subdivided into several smaller dose increments using the PreciseInhale (data collected from inhalation sessions No. 3 and 4). Outcome measured in session 3-4
Air flow rate | Collected during inhalation session, approx. for 5 min
  Measure air flow rates and aerosol concentration- and timing in the ventilation manoeuvre to demonstrate that regional targeting can be achieved with PreciseInhale bolus-breath hold method (data collected from inhalation sessions No 3 and 4). Outcome measured in session 3-4
Aerosol concentration | Collected during inhalation session, approx. for 5 min
  Measure air flow rates and aerosol concentration- and timing in the ventilation manoeuvre to demonstrate that regional targeting can be achieved with PreciseInhale bolus-breath hold method (data collected from inhalation sessions No 3 and 4). Outcome measured in session 3-4.
Acutal bolus volume | Collected during inhalation session, approx. for 5 min
  Measure air flow rates and aerosol concentration- and timing in the ventilation manoeuvre to demonstrate that regional targeting can be achieved with PreciseInhale bolus-breath hold method (data collected from inhalation sessions No 3 and 4). Outcome measured in session 3-4.
Chase air volume | Collected during inhalation session, approx. for 5 min
  Measure air flow rates and aerosol concentration- and timing in the ventilation manoeuvre to demonstrate that regional targeting can be achieved with PreciseInhale bolus-breath hold method (data collected from inhalation sessions No 3 and 4). Outcome measured in session 3-4.
Actual number of inhalations | Collected during inhalation session, approx. for 5 min
  Measure air flow rates and aerosol concentration- and timing in the ventilation manoeuvre to demonstrate that regional targeting can be achieved with PreciseInhale bolus-breath hold method (data collected from inhalation sessions No 3 and 4). Outcome measured in session 3-4.
Correlation between two outcomes: AUC (weight-adjusted) -inhaled/exhaled dose | AUC from pre-dose to up to 24 hours post-dose. Inhaled/exhaled dose collected post-dose at one occasion.
  Area under the curve from time 0 to time t adjusted for weight and correlated to inhaled/exhaled dose. Outcome measured in session 2-4.

SECONDARY OUTCOMES:
Adverse events (AEs) | From start of first inhalation training until the end-of- study visit, an average of 5 weeks.
  Frequency, intensity and seriousness of adverse events (AEs). The intensity grades were defined as mild, moderate and severe. AEs were assessed as not related, possibly or probably related to the investigational device, the procedures or the test drug substances according to MDCG 2020-10/1. Outcome measured in session 1-4.
Device deficiencies (DD) | From start of first inhalation training until the end-of- study visit, an average of 5 weeks
  Frequency and nature of device deficiencies (DD). A device deficiency (DD) is defined as any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors, or inadequacy in information supplied by the manufacturer. If a DD is assessed by the Investigator or the CTC's Pharmacovigilance department (CTC PV), as an event that could have led to an SAE if appropriate action not taken, intervention not made or circumstances less fortunate the event is to be reported as a reportable event. For registration of action taken with the device the following definitions will be used: removal, discarded, quarantined and treatment withdrawn. Outcome measured in session 1-4.
Number of changes in vital signs judged as clinically significant by Principal Investigator | Vital signs will be checked at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 6 weeks
  Systolic and diastolic blood pressure and pulse will be measured in supine position after 10 minutes of rest. Outcome measured in session 1-4.
Number of changes in electrocardiogram (ECG) judged as clinically significant by Principal Investigator | ECG will be checked at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 6 weeks
  Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. Heart rate and PQ/PR, QRS, QT and QTcF intervals will be recorded. Outcome measured in session 1-4.
Number of changes in safety laboratory parameters judged as clinically significant by Principal Investigator | Blood samples will be collected at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 6 weeks
  Blood samples for analysis of clinical chemistry and haematology parameters will be collected and sent to the certified clinical chemistry laboratory at Uppsala University Hospital and analysed by routine analytical methods. Urinalysis will be performed at the research clinic using dip sticks. Outcome measured in session 1-4.
Number of changes in physical examination judged as clinically significant by Principal Investigator | Physical examination will be performed at pre-defined timepoints from the screening visit until the end-of- study visit, an average of 6 weeks
  A complete physical examination included assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. Outcome measured in session 1-4.
Device user experience questionnaire completed by PreciseInhale operator | Completed once after treatment period 4 (visit 8), approximately 15 min
  A device user experience questionnaire will be completed by the PreciseInhale operator after completion of last inhalation session with the PreciseInhale. Answers will be entered in the eCRF by the study personnel. Outcome measured after session 4 but operator experience from session 2-4 collected.
Device user experience questionnaire completed by study subject | Completed once after treatment period 4 (visit 8), approximately 15 min
  A device user experience questionnaire will be completed by the study subject after completion of last inhalation session with the PreciseInhale. Answers will be entered in the electronic patient reported outcomes (ePRO) system ViedocMe by the study subjects. Outcome measured after session 4 but subject experience from session 2-4 collected.

CONTACTS AND LOCATIONS:
Overall Officials: Manoush Masarrat, Study Chair — Inhalation Sciences AB
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No